CLINICAL TRIAL: NCT06717321
Title: Percutaneous Endoscopic Gastrostomy Versus Percutaneous Endoscopic Gastrostomy With Jejunal Extension: A Randomized Clinical Trial
Brief Title: Percutaneous Endoscopic Gastrostomy Versus Percutaneous Endoscopic Gastrostomy With Jejunal Extension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty Enrolling
Sponsor: Jerry Dang (Other)
Responsible Party: Sponsor-Investigator, Jerry Dang, Associate Professor of Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-170
Record Dates: First submitted 2024-12-03; First posted 2024-12-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Aspiration Pneumonias; Tube Feeding; Enteral Feeds
Keywords: tube feeds; aspiration pneumonia; peg; peg-J; enteral feeding
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG arm: Patients receiving the 20-French pull-type PEG tube (Active Comparator): PEG Arm:
  Participants receive a 20-French pull-type percutaneous endoscopic gastrostomy tube placed into the stomach using standard safe track technique with transillumination and 1:1 finger indentation. The tube is positioned midway between the greater and lesser curves of the stomach. Continuous tube feeds begin 24 hours after placement. Follow-up period is 30 days.
  Interventions: Procedure: (Arm 1): PEG
- PEG-J arm: Patients receiving the 24-French pull-type PEG with 12-French jejunal extension tube (Active Comparator): Participants receive a 24-French pull-type percutaneous endoscopic gastrostomy tube with a 12-French jejunal extension. After standard PEG placement, the jejunal extension tube is advanced past the pylorus and secured to the small bowel wall with endoclips as indicated. Continuous tube feeds begin 24 hours after placement. Follow-up period is 30 days.
  Interventions: Procedure: (Arm 2): PEG-J

INTERVENTIONS:
Procedure: (Arm 1): PEG — A 20-French pull type percutaneous endoscopic feeding tube placed into the stomach using endoscopic guidance
  Arms: PEG arm: Patients receiving the 20-French pull-type PEG tube
Procedure: (Arm 2): PEG-J — 24-French pull type percutaneous endoscopic feeding tube placed into the stomach with a 12-French jejunal extension tube advanced through the PEG and positioned post-pyloric in the small bowel using endoscopic guidance
  Arms: PEG-J arm: Patients receiving the 24-French pull-type PEG with 12-French jejunal extension tube

SUMMARY:
The goal of this clinical trial is to learn if placing a feeding tube with a small bowel extension (called Percutaneous Endoscopic Gastrostomy With Jejunal Extension [PEG-J]) is better at preventing pneumonia than a standard feeding tube (called Percutaneous Endoscopic Gastrostomy [PEG]) in people who need long-term tube feeding. Researchers want to know if people who receive a PEG-J have fewer cases of pneumonia in the first 30 days compared to those who receive a standard PEG, and whether PEG-J tubes require more follow-up procedures to fix tube problems.

Researchers will compare two different types of feeding tubes: a standard feeding tube that goes into the stomach (PEG) versus a feeding tube that extends past the stomach into the small intestine (PEG-J). This will help determine which type of feeding tube is safer and works better for patients.

Participants will be randomly assigned to receive either a PEG or PEG-J feeding tube through a minimally invasive procedure. They will start receiving nutrition through the tube 24 hours after placement and be monitored for 30 days to check for problems like pneumonia or tube malfunction, while receiving regular medical care from their treating doctors.

The study is open to people who are 18 years or older and need a new feeding tube for long-term nutrition. People cannot take part if they have pneumonia, COVID-19, an existing feeding tube, previous stomach surgery, gastroparesis (a condition affecting stomach movement), digestive system blockage, are pregnant, or are in prison. All participants must understand English.

Participation is voluntary, and participants can leave the study at any time. The study team will carefully monitor all participants for any problems throughout the 30-day period

DETAILED DESCRIPTION:
This randomized clinical trial investigates the comparative efficacy of percutaneous endoscopic gastrostomy (PEG) versus percutaneous endoscopic gastrostomy with jejunal extension (PEGJ) for long-term enteral access. The study addresses a critical knowledge gap in the literature regarding the optimal approach for enteral feeding in patients at risk for aspiration.

Current evidence suggests that aspiration pneumonia occurs in up to 30% of patients following PEG placement, with some studies demonstrating aspiration in up to 38% of patients immediately after enteral feeding administration. This high rate is hypothesized to result from gastric reflux. While PEGJ has been proposed as a potential solution by advancing feeds beyond the pylorus, existing evidence consists primarily of small case series and retrospective studies, with reported aspiration pneumonia rates of approximately 10%. However, the methodological limitations of these studies and contradicting findings create uncertainty about the optimal approach.

A recent meta-analysis of enteral feeding in critically ill patients suggested potential benefits of post-pyloric feeding, but included moderate to low quality evidence and did not directly compare PEG versus PEGJ. Furthermore, some researchers argue that aspiration events may result from oropharyngeal dysphagia rather than gastric reflux, potentially limiting the benefit of jejunal extension.

The study employs a prospective, randomized design with 1:1 allocation using distance randomization via RedCap to ensure allocation concealment. Sample size calculation was based on detecting a 20% difference between groups in aspiration pneumonia rates, with power analysis accounting for a statistical power of 0.8 using chi-square test methodology.

The technical aspects of tube placement follow standardized protocols. For PEG placement, a 20-French pull-type tube is positioned using safe track technique with transillumination and 1:1 finger indentation, placing the tube midway between the greater and lesser curves of the stomach. The PEGJ procedure begins similarly but utilizes a 24-French pull-type PEG followed by advancement of a 12-French jejunal extension tube, which is secured to the small bowel wall with endoclips as indicated.

Both groups will receive continuous feeding rather than bolus feeding to standardize the feeding methodology. The study design accounts for potential confounding factors by excluding patients with conditions that might independently affect aspiration risk or tube function, such as gastroparesis or prior upper gastrointestinal surgery.

The research addresses both clinical efficacy and practical considerations, as PEGJ tubes have reported malfunction rates of up to 50%, potentially requiring additional interventions. This prospective investigation will provide high-quality evidence to guide clinical decision-making, balancing the potential benefits of aspiration reduction against the risks of tube dysfunction and need for reintervention.

Statistical analysis will be conducted by an internal biostatistician using appropriate methodologies for both continuous and categorical variables, with adjustments for non-normal distributions when necessary. The study's 30-day follow-up period was selected based on typical timeframes for post-procedure complications and tube-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Requires feeding access as determined by treating provider

Exclusion Criteria:

* Concurrent pneumonia at time of enrollment
* Concurrent COVID-19 diagnosis
* Prior feeding access (transabdominal feeding access)
* Prior upper gastrointestinal surgery (previous gastric resection surgery)
* Gastroparesis
* Obstruction or pseudo-obstruction
* Pregnancy
* Contraindication to undergo upper endoscopy
* Prisoners
* Primary language is not English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Developed Post-Procedure Pneumonia | From day of procedure (day 0) through 30 days post-procedure
  Diagnosis of pneumonia will be determined based on clinical judgment of the treating provider and must be explicitly documented as "pneumonia" in the medical record.

SECONDARY OUTCOMES:
Number of Participants Requiring Additional Procedures Due to Tube Malfunction | From day of procedure (day 0) through 30 days post-procedure
  A tube malfunction is defined as any issue requiring an additional procedure to maintain tube function.
Number of Participants with Post-Operative Complications | From day of procedure (day 0) through 30 days post-procedure
  Any documented post-operative complication will be counted, including but not limited to bleeding, infection, and injury to organs or structures
Total Procedure Time in Minutes from Start to Completion of Feeding Tube Placement | Day of procedure
  Measurement of total operative time from the start of the endoscopic procedure until completion of feeding tube placement and final endoscopic verification of proper positioning. Time will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Dang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Based on the protocol's data collection and privacy sections, individual participant data (IPD) that underlie the results reported in published articles will not be shared. The IRB-approved protocol specifies that data access is restricted to the research team and regulatory instances at Cleveland Clinic. As per protocol's privacy and confidentiality section, data will be safeguarded in REDCap with access limited to authorized study personnel, and data retention is specified for 5 years after study completion. These limitations on data sharing are in place to maintain participant confidentiality and comply with the privacy protections promised during the informed consent process.

REFERENCES:
- [Background] Fox KA, Mularski RA, Sarfati MR, Brooks ME, Warneke JA, Hunter GC, Rappaport WD. Aspiration pneumonia following surgically placed feeding tubes. Am J Surg. 1995 Dec;170(6):564-6; discussion 566-7. doi: 10.1016/s0002-9610(99)80016-6. PMID 7492001
- [Background] Chang WK, Huang HH, Lin HH, Tsai CL. Evaluation of Oropharyngeal Dysphagia in Patients Who Underwent Percutaneous Endoscopic Gastrostomy: Stratification Risk of Pneumonia. JPEN J Parenter Enteral Nutr. 2020 Feb;44(2):239-245. doi: 10.1002/jpen.1592. Epub 2019 Apr 14. PMID 30983013
- [Background] Gauderer MW, Ponsky JL, Izant RJ Jr. Gastrostomy without laparotomy: a percutaneous endoscopic technique. J Pediatr Surg. 1980 Dec;15(6):872-5. doi: 10.1016/s0022-3468(80)80296-x. PMID 6780678
- [Background] Minard G. The history of surgically placed feeding tubes. Nutr Clin Pract. 2006 Dec;21(6):626-33. doi: 10.1177/0115426506021006626. PMID 17119170
- [Background] Seres DS, Valcarcel M, Guillaume A. Advantages of enteral nutrition over parenteral nutrition. Therap Adv Gastroenterol. 2013 Mar;6(2):157-67. doi: 10.1177/1756283X12467564. PMID 23503324
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056